CLINICAL TRIAL: NCT06050720
Title: An Exploratory Study of a Novel, Low-cost Sleep Apnoea Screening Device to Compare Its Capability to Identify Apnoeas and Hypopneas With Current Standard Sleep Apnoea Test Devices
Brief Title: Sleep Apnoea Breathing Record Exploratory Study (SABRES)
Acronym: SABRES
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospitals of North Midlands NHS Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 3282
Record Dates: First submitted 2023-09-06; First posted 2023-09-22 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Participants will have been referred to the sleep clinic at Royal Stoke Hospital for a diagnosis of a possible sleep disorder, possibly sleep apnoea. If they enrol in the study the participants will be asked to wear the Apne-Scan DC1 device to changing pressures in the user's breathing whilst asleep.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sleep disorder patients (Other): The study participants have been referred by a clinician to the sleep clinic for diagnosis of a sleep disorder, possibly sleep apnoea.
  Interventions: Device: Apne-Scan DC1 device

INTERVENTIONS:
Device: Apne-Scan DC1 device — The primary objective of this exploratory study is to assess Apnea-Tech's UKCA Class I Apne-Scan DC1 sleep apnoea screening device in assisting a clinical diagnosis of sleep apnoea in comparison to standard sleep apnoea test devices (ResMed NOX T3 and Phillips Alice Night One).

SUMMARY:
During sleep, many people have times when they breathe shallowly or completely stop. If a person stops breathing for more than 10 seconds, this is called an 'apnoea'. If shallow breathing lasts for more than 10 seconds, it is called a 'hypopnoea'. If a person has these events frequently, it disrupts their sleep and they do not awake refreshed. It can also put strain on the heart, leading to cardiovascular conditions. These sleep disorders, usually called 'Sleep Apnoea', can be treated for most people using 'continuous positive airways pressure', CPAP. Current tests for sleep apnoea, usually used at home, are expensive, complicated for patients to use and do not monitor actual breathing. The new test, called Apne-Scan, is very simple and will cost less than the standard tests. It just requires the user to wear a mask, similar to ones used for CPAP treatment, overnight and then send the mask off for data analysis. The Apne-Scan mask, developed with taxpayer funding, is fitted with a pressure sensor to monitor actual breathing. People between the ages of 18-70 who have been referred to the sleep clinic at Royal Stoke University Hospital are eligible to participate in this exploratory study. They will wear the Apne-Scan mask at the same time as their standard overnight sleep apnoea test. The breathing data collected by Apne-Scan will be analysed by Apnea-Tech Limited, the device manufacturers, so that it can be compared to the data captured by the standard sleep apnoea test.

ELIGIBILITY:
Inclusion Criteria:

* Have been referred by a clinician to the sleep clinic for diagnosis of a sleep disorder, possibly sleep apnoea.
* Be about to be screened for possible sleep apnoea using a standard sleep apnoea test device.
* Be between the ages of 18 and 75 and have provided informed consent for the study

Exclusion Criteria:

* Have not been referred by a clinician to a sleep clinic for diagnostic tests for sleep disorders other than for possible sleep apnoea.
* Cannot tolerate wearing a mask overnight.
* Cannot remove a mask should they become distressed.
* Are not capable of understanding the English language version of Apne-Scan's Instructions For Use (IFU).
* Are under the age of 18 years old or over the age of 75 years old.
* Are not capable of giving informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Breathing pressure changes | 2 months
  The primary outcome of interest is the data capture of the changing pressures in the user's breathing, whilst asleep, as recorded by the Apne-Scan DC1 device

SECONDARY OUTCOMES:
Comparison between sleep apnoea devices | 2 months
  An overall comparison of the sleep apnoea screening output from Apne-Scan DC1 with that from standard sleep apnoea test devices (ResMed NOX T3 and Phillips Alice Night One).
Severity of sleep apnoea | 2 months
  A comparison stratified by the severity of the sleep apnoea indicated by standard sleep apnoea test devices.
Severity of hypopnoea | 2 months
  A comparison stratified by the severity of the hypopnoea indicated by standard sleep apnoea test devices.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of North Midlands NHS Trust, Stoke-on-Trent, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No identifiable data will be used in the results of the study